CLINICAL TRIAL: NCT04334330
Title: Palbociclib, Trastuzumab, Pyrotinib and Fulvestrant Treatment in Patients With Brain Metastasis From ER/PR Positive, HER-2 Positive Breast Cancer: A Multi-center, Prospective Study in China
Brief Title: Palbociclib, Trastuzumab,Pyrotinib and Fulvestrant Treatment in Patients With Brain Metastasis From ER/PR Positive, HER-2 Positive Breast Cancer: A Multi-center, Prospective Study in China
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, wang shusen, Chief Physician, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCBCS025
Record Dates: First submitted 2020-04-02; First posted 2020-04-06 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Breast Cancer; Brain Metastases
Keywords: breast cancer, brain metastasis, Palbociclib, CDK4/6 inhibitor, pyrotinib, fulvestrant, trastuzumab, HER2-positive, ER/PR positive, hormonal receptor positive
MeSH Terms: conditions — Breast Neoplasms; Brain Neoplasms | interventions — palbociclib; Trastuzumab; pyrotinib; Fulvestrant

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental)
  Interventions: Drug: Palbociclib, Trastuzumab, Pyrotinib and Fulvestrant

INTERVENTIONS:
Drug: Palbociclib, Trastuzumab, Pyrotinib and Fulvestrant — ER/PR positive, HER2-positive breast cancer patients with brain metastatic lesions receive palbociclib PO daily on days 1-21, combined with trastuzumab IV every three weeks, pyrotinib PO daily and fulvestrant IM every 4 weeks. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

SUMMARY:
The objective of this study is to evaluate the efficacy of combination of palbociclib, trastuzumab and pyrotinib with fulvestrant in ER/PR positive and HER2-positive breast cancer patients with brain metastasis.

ELIGIBILITY:
Inclusion Criteria

1. Age greater than 18 years old
2. Female patients aged 18 years or older
3. Histologically confirmed ER/PR positive, HER2-positive metastatic breast cancer (ER/PR≥1% by IHC; HER-2 3+ by immunohistochemistry (IHC); if IHC score of 2, fluorescence in situ hybridization (FISH) ratio must be greater than 2.0; if FISH less than 2.0, HER2 copy number must be greater than 6; NOTE: Brain lesions are not required to have pathologic confirmation)
4. Patients must have a life expectancy of at least 12 weeks at the time of registration
5. Eastern Cooperative Oncology Group (ECOG) performance status >= 2
6. Measurable disease in the brain, defined as at least 1 lesion measuring >= 10 mm on MRI at the time of registration
7. If patients are on corticosteroids, they must have been on a stable or decreasing dose >= 5 days prior to obtaining their baseline gadolinium (Gd)-magnetic resonance imaging (MRI) of brain; this MRI is to be obtained within 28 days of registration; NOTE: If patient needs escalation of steroids prior to therapy, or are on unstable doses of steroids they are not eligible
8. Patients who have a history of hypersensitivity reaction to one of the compounds or incorporated substances used in this protocol; AND/OR patients who have had prior exposure to fulvestrant, everolimus, pyrotinib or CDK4/6 inhibitors and had a disease progression during treatment are not eligible.
9. Patients must not have received systemic therapy within 2 weeks of initiating palbociclib; NOTE: For patients on trastuzumab, they can remain on the drug; no break or washout period required
10. Patients must exhibit adequate bone marrow, liver, and renal function, within 14 days prior to registration, defined as:
11. Absolute neutrophil count (ANC) >= 1,000/mm^3 (growth factor support is permitted)
12. Platelets >= 50,000/mm^3 (may be reached by transfusion)
13. Hemoglobin >= 10 gm/dl (may be reached by transfusion)
14. Glutamate pyruvate transaminase (GPT)/glutamate oxaloacetate transaminase (GOT) < 3 x upper limit of normal (ULN) (or < 5 x ULN in case of liver metastasis)
15. Bilirubin < 3 x ULN (or < 5 x ULN in case of liver metastasis)
16. Creatinine < 1.5 x ULN
17. Women of childbearing age must have a serum pregnancy test within 7 days before enrollment, and the result should be negative, and are willing to use a medically recognized high-efficiency contraceptive during the study period and within 1 year after the last administration of the study drug.
18. Has not undergone a hysterectomy or bilateral oophorectomy
19. Has had menses at any time in the preceding 12 consecutive months (and therefore has not been naturally postmenopausal for > 12 months)
20. Female patients must have a negative urine pregnancy test within 7 days prior to registration; if urine test is positive, it should be followed by serum pregnancy test
21. Patients must sign an informed consent prior to registration and before undergoing any study-specific procedures indicating that they are aware of the investigational nature of this study
22. Patient must have the ability to comply with all study requirements

Exclusion Criteria

1. Any uncontrolled neurological symptom attributed to CNS metastasis
2. Brain metastasis must not be impending herniation or other significant vasogenic edema requiring increasing steroid doses; lesions must not have frank hemorrhage
3. Patients with leptomeningeal disease are not eligible for participation
4. Patients have been treated with WBRT. The selected intracranial target lesion has received local treatment (surgical resection or SRS). Acute effects related to surgery or SRS have not recover
5. Any significant medical illnesses or infection that, in the investigator's opinion, cannot be adequately controlled with appropriate therapy or would compromise the patient's ability to tolerate this therapy are not eligible for participation
6. Known human immunodeficiency virus (HIV) positive status
7. Known active hepatitis B and/or C
8. Patients who have a history of hypersensitivity reaction to one of the compounds or incorporated substances used in this protocol; AND/OR patients who have had prior exposure to compounds of similar chemical or biologic composition to palbociclib or lapatinibpyrotinib and PD during treatment are not eligible.
9. Patients being treated with any other experimental agents/clinical trials are not eligible for participation; if the patient is on any investigational agent, a wash-out period of minimum 2 weeks prior to registration is mandatory for the patient to be eligible for the study
10. Inability to swallow capsules, malabsorption syndrome or gastrointestinal disease that severely affects the absorption of study drugs, major resection of the stomach or small bowel, or gastric bypass procedure
11. Patients who have an uncontrolled intercurrent illness including, but not limited to any of the following, are not eligible:
12. Ongoing or active infection requiring systemic treatment
13. Symptomatic congestive heart failure
14. Unstable angina pectoris
15. Cardiac arrhythmia: except atrial fibrillation (AF) and supraventricular tachycardia (SVT) that are controlled by medication
16. Psychiatric illness/social situations that would limit compliance with study requirements
17. Any other illness or condition that the treating investigator feels would interfere with study compliance or would compromise the patient's safety or study endpoints

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2020-12-04 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate in the CNS | Up to 3 years
  Assess the response rate in the CNS by MRI according to modified Response Assessment in modified RECIST 1.1 criteria. Objective CNS response is defined as at least 30% decrease in the sum of diameters of CNS target lesions in the absence of new lesions (defined as ≥ 6 mm), increased steroid use, progressive neurological symptoms, and progressive extra-CNS disease as assessed by RECIST 1.1. Confirmatory scans are not required.

SECONDARY OUTCOMES:
Overall Survival | Up to 3 years
  OS is defined as the time from treatment initiation until death due to any cause
Progression Free Survival | Up to 3 years
  PFS is defined as the time from treatment initiation to documented disease progression
Overall Response Rate | Up to 3 years
  Evaluate systemic ORR defined as partial response or complete response assessed by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
Time to CNS progression | Up to 3 years
  Time to CNS progression will be defined as the time from treatment initiation to documented disease progression (modified RECIST 1.1 criteria) in the CNS
Time to radiotherapy | Up to 3 years
  Time to radiotherapy is defined as the time from the date of inclusion to the date of event defined as the initiation of radiotherapy

OTHER OUTCOMES:
Change in quality of life in patients receiving study drug combination | At baseline, 2 months and 4 months
  Quality of life measures will be assessed at baseline, 2 months and 4 and will be collected using patient reported outcome questionnaires: Functional Assessment of Cancer Therapy-Brain (FACT-Br), EORTC QLQ-BR23

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Shusen Wang, Guangzhou, Guangdong
  - State Key Laboratory of Oncology in South China, Sun Yat-sen University Cancer Center, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chen D, Xu F, Lu Y, Xia W, Du C, Xiong D, Song D, Shi Y, Yuan Z, Zheng Q, Jiang K, An X, Xue C, Huang J, Bi X, Chen M, Zhang J, Wang S, Hong R. Pyrotinib and trastuzumab plus palbociclib and fulvestrant in HR+/HER2+ breast cancer patients with brain metastasis. NPJ Breast Cancer. 2024 Jun 13;10(1):45. doi: 10.1038/s41523-024-00646-2. PMID 38871705